CLINICAL TRIAL: NCT02796599
Title: Impact of Various Interfaces of Non-invasive Ventilation on Performance During Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Interfaces of Non-invasive Ventilation on Performance in Patients With Chronic Obstructive Pulmonary Disease
Acronym: Exercise-NIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Exercise-NIV
Record Dates: First submitted 2016-05-30; First posted 2016-06-10 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Non Invasive Ventilation; Exercise, Aerobic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

ARMS (2):
- CWLT with facial mask (Experimental): This study has a cross-over design. Patients will achieve CWLT with non-invasive ventilation using facial or nasal mask in a randomised order.
  Interventions: Device: Non invasive ventilation during exercise with facial or nasal mask.
- CWLT with nasal mask (Experimental): This study has a cross-over design. Patients will achieve CWLT with non-invasive ventilation using facial or nasal mask in a randomised order.
  Interventions: Device: Non invasive ventilation during exercise with facial or nasal mask.

INTERVENTIONS:
Device: Non invasive ventilation during exercise with facial or nasal mask. — Every patients will achieve 3 constant work load test (CWLT) at 75% Wpic. The first CWLT will be realized without any ventilatory support. The 2 others CWLT will be achieved with non-invasive ventilation support using facial or nasal interface in a randomized order.

SUMMARY:
The purpose of this study is to determine wether the interface (facial or nasal mask) influences performance in patients with chronic obstructive pulmonary disease exercising with non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chronic obstructive pulmonary disease Gold III-IV
* Eligible for pulmonary rehabilitation
* Exercise limitation : at least respiratory limitation (ventilatory reserve ≤ 30%)

Non-inclusion Criteria:

* Pregnant woman or likely to be
* Familiar with home non-invasive ventilation
* Patient under guardianship

Exclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Endurance time (Tlim, in second) during Constant Work Load Test (CWLT). | The outcome will be measure after every CWLT. The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Patients will achieve 3 Constant Work Load Test Under different conditions (1 without noninvasive ventilation and 2 with noninvasive ventilation using in a randomised order facial or nasal mask). Endurance time (sec) will be recorded at the end of every test.

SECONDARY OUTCOMES:
Comfort of different masks using numerical scale (0-10) after exercising with noninvasive ventilation. | The outcome will be measure after every CWLT achieved with noninvasive ventilation. CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  The comfort of the different interfaces is assessed after every CWLT using numerical scale.
Dyspnea during CWLT using modified Borg Scale (0-10). | The outcome will be measure during every CWLT.The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be collected every 30s during tests.
  The dyspnea will be assessed every 30sec during CWLT. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Exhaustion during CWLT using modified Borg Scale (0-10). | The outcome will be measure during every CWLT.The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be collected every 30s during tests.
  The exhaustion will be assessed every 30sec during CWLT. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Heart rate (rpm) during CWLT using capnograph. | The outcome will be measure during every CWLT (with or without noninvasive ventilation).The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Blood pressure (mmHg) before and after every CWLT using electrical blood pressure device. | The outcome will be assessed before and after every CWLT. The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
Oxygen saturation (SpO2, %) during CWLT using capnograph. | The outcome will be measure during every CWLT (with or without noninvasive ventilation).The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Transcutaneous carbon dioxide pressure (PtcCO2, mmHg) during CWLT using capnograph. | The outcome will be measure during every CWLT (with or without noninvasive ventilation).The 3 CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Respiratory rate (rpm) during CWLT with noninvasive ventilation using ventilator monitoring. | The outcome will be measure during CWLT with noninvasive ventilation. CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 2 tests) and iso time (defined as the Tlim or the shortest test).
Inspiratory tidal volume (Vti, in liter) during CWLT with noninvasive ventilation using ventilator monitoring. | The outcome will be measure during CWLT with noninvasive ventilation. CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 2 tests) and iso time (defined as the Tlim or the shortest test).
Leak (liter per minute) during CWLT with noninvasive ventilation using ventilator monitoring. | The outcome will be measure during CWLT with noninvasive ventilation. CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 2 tests) and iso time (defined as the Tlim or the shortest test).

OTHER OUTCOMES:
Ventilatory asynchronism during CWLT with noninvasive ventilation using ventilator monitoring. | The outcome will be measure during CWLT with noninvasive ventilation. CWLT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Outcome will be continuously recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Viacroze, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Catherine Tardif, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; David Debeaumont, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Tristan Bonnevie, PT, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France
Locations (1):
- ADIR Association, Bois-Guillaume, France